CLINICAL TRIAL: NCT05680298
Title: Open-label Exploratory Study to Evaluate the Effect of Dupilumab on Skin Barrier Function in Chinese Pediatric Patients With Moderate-to-severe Atopic Dermatitis
Brief Title: Dupilumab-pediatric Skin Barrier Function and Lipidomics Study in Patients With Atopic Dermatitis in China
Acronym: PELISTAD CN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LPS17244; U1111-1272-6639 (Registry Identifier: ICTRP); 2024-000402-15 (EudraCT Number)
Record Dates: First submitted 2022-12-26; First posted 2023-01-11 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AD patients (Experimental): Pediatric patients (≥6 and <12 years of age) with moderate-to-severe AD will receive a SC injection of dupilumab depending on the body weight
  Interventions: Drug: Dupilumab
- Healthy volunteers (No Intervention): Except for IMPs administration, skin barrier function assessments for healthy volunteers are conducted at the same time and in the same measurement conditions as for AD patients.

INTERVENTIONS:
Drug: Dupilumab — solution for injection, Subcutaneous injection
  Other Names: Dupixent
  Arms: AD patients

SUMMARY:
This is a 32-week, open-label, exploratory study with a 4-week screening period, 16-week treatment phase designed to investigate dupilumab's effect on skin barrier function as measured by TEWL before and after STS in approximately 20 pediatric patients with moderate-to-severe AD (not more than 24 patients aged ≥6 and <12 years old), and a 12-week follow-up period. Patients will have 1 on-site visit/week, up to Week 4, 1 on-site visit every 2 weeks from Week 4 to Week 8, and 1 on-site visit every 4 weeks from Week 8 to Week 16 End of Treatment (EoT) phase visit, and every 6-weeks thereafter during the follow-up period and by this will end the study for each participant (End of Study [EoS]). The maximum duration of the study per participant will be 32 weeks (including screening period).

Skin barrier function in approximately 10 healthy volunteers (not more than 20 healthy participants aged ≥6 and <12 years old) matched for age (match on age ±2 years), gender, location of targeted lesion area, and study site to the AD cases will be assessed in a similar manner at baseline, and will have 1 on-site visit/week, up to Week 4, 1 on-site visit every 2 weeks from Week 4 to Week 8, and 1 on-site visit every 4 weeks from Week 8 to Week 16 EoT phase visit, and every 6-weeks thereafter during the follow-up period, serving as a reference comparator for skin barrier function.

DETAILED DESCRIPTION:
32 weeks

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for AD patients

* Participant must be between ≥6 to <12 years of age inclusive, at the time of signing the informed consent.
* Male or female.
* Patients with AD diagnosis according to Hanifin and Rajka criteria at least 1 year before screening.
* Investigator Global Assessment score of ≥3 (for US patients) or IGA ≥4 (for EU patients) at screening (on the 0 to 4 scale) depending on approved label indication in the country.
* Patients with moderate-to-severe AD are eligible to be treated with dupilumab according to product label.
* Patients with AD must have active lesions on the upper limbs or lower limbs (including trunk, if needed), with severity for lesion erythema or edema/papulation ≥2 at screening on the 0 to 3 scale of the ISS.
* Participants should have a non-lesional (normal looking) skin area 4 cm from the edge of the lesional area. If unable to identify non-lesional skin 4 cm from the lesional area, it is acceptable to identify normal looking skin as close to the lesion as possible.
* Willing to refrain from applying any topical medications on the target assessment areas (including lesional and non-lesional) throughout the study until EoS unless necessary to alleviate intolerable symptoms.
* Willing to refrain from showers or soak in a bathtub with soaps and body washes within 6 hours before TEWL assessments.
* Willing to NOT apply any moisturizers to the areas of the skin that are targeted assessment areas (lesional and non-lesional) during the entire study from Day -7 to Week 28 (EoS).
* Willing and able to comply with all clinic visits and study-related procedures.
* 15 kg ≤ body weight <60 kg

Inclusion Criteria for HEALTHY VOLUNTEERS

* Age and gender matched (match on age ±2 years) to a selected AD patient by study site.
* No current dermatologic or systemic condition that could interfere with the assessments.
* 15 kg ≤ body weight <60 kg
* Male or female - - - -

Exclusion Criteria:

Medical conditions

* Previous treatment with dupilumab within 6 months prior to screening.
* Skin conditions other than AD that can confound assessments in the area of TEWL assessments in the opinion of the Investigator (ie, skin atrophy, ichthyosis, tinea infection, contact dermatitis).
* Cracked, crusted, oozing, or bleeding AD lesions in the designated lesional assessment area leaving insufficient skin that is adequate for TEWL assessments.
* Hypersensitivity to the active substance or to any of the excipients of dupilumab.
* Ocular disorder that in the opinion of the Investigator could adversely affect the individual's risk for study participation.
* Systemic AD treatment, cyclosporine A (CsA), systemic corticosteroids, azathioprine (AZA), methotrexate (MTX), mycophenolate mofetil (MMF), or Janus kinase (JAK) inhibitors or phototherapy within 4 weeks of baseline.
* Topical AD treatment within 1 week of baseline. Face and neck may be treated with topical steroids during the washout period if approved by the Investigator.
* Severe concomitant illness(es) that, in the Investigator's judgment, would adversely affect the patient's participation in the study.
* History of hypersensitivity reaction to tape or adhesives used in desquamme discs.
* Patients administered live attenuated vaccines within the 4 weeks prior to the baseline visit or need to receive live (attenuated) vaccinations through Week 28.

Prior/concomitant therapy

* Treatment with an investigational medication within 16 weeks or within 5 half-lives (if known) prior to Day 1, whichever is longer.
* Patients who received a live vaccine within 4 weeks of baseline.

Prior/concurrent clinical study experience

- Current participation in another investigational or interventional clinical study

Other exclusions

* Planned or anticipated major surgical procedure during the patient's participation in this study.
* Healthy volunteers with a personal history of an atopic condition.
* Healthy volunteers with use of any topical treatment anywhere except Cetaphil®, Vanicream™, E45 cream or the preferred moisturizer not containing additives on non-targeted skin areas.
* Female of childbearing potential* and sexually active, who is unwilling to use highly effective methods of contraception prior to the initial dose, during the study and for at least 120 days after the last dose of study drug.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in TEWL after 5 STS assessed on lesional skin at Week 16 in AD patients. | From baseline to week16

SECONDARY OUTCOMES:
Change from baseline in TEWL before and after 10, 15, 20 STS assessed on lesional skin in AD patients at Week 16. | From baseline to week16

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Beijing Children's hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: LPS17244 Plain language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25296&tenant=MT_SNY_9011